CLINICAL TRIAL: NCT06753812
Title: Investigation of the Effect of Constraint Induced Movement Therapy Applied to the Lower Extremity on Balance, Gait and Lower Extremity Functions in Individuals With Unilateral Cerebral Palsy
Brief Title: Investigation of the Effect of Constraint Induced Movement Therapy Applied to the Lower Extremity on Lower Extremity Functions in Individuals With Unilateral Cerebral Palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ayşe Neriman NARİN, Assistant Professor, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-ANN-02
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy Spastic Hemiplegic
Keywords: cerebral palsy; Surface Electromiyography; lower extremity
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups with a conventional therapy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint induced movement therapy group (Active Comparator): Children in this group will receive constraint induced movement therapy in addition to conventional physical therapy twice a week.
  Interventions: Other: constraint induced movement therapy
- Control group (Other): Children in this group will continue to receive their treatment twice a week at the special education and rehabilitation center where they are currently registered and attending.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: constraint induced movement therapy — Children in this group will receive constraint induced movement therapy for 10 sessions over 2 weeks, each session lasting 90 minutes, in addition to the treatment they receive 2 days a week at the special education and rehabilitation centers they attend.
  Arms: Constraint induced movement therapy group
Other: Control (Standard treatment) — Children in this group will continue to receive their treatment at the special education and rehabilitation center they attend, two days a week for 40 minutes.
  Arms: Control group

SUMMARY:
Lower extremity constraint induced movement therapy has been applied to individuals with multiple sclerosis, stroke, subacute and chronic hemiparesis in recent years and positive results have been reported. However, there is no study in the literature regarding the application of this treatment method to the pediatric population. In order to address this gap in the literature, we planned to conduct this study to examine the possible effects of lower extremity constraint induced movement therapy on lower extremity functions, balance and gait parameters in individuals with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is an umbrella term covering a group of non-progressive motor disorder syndromes secondary to lesions or anomalies in the immature brain. The global prevalence of CP is 1.5-3.8 per 1000 births. The most common problems in CP are motor disorders such as spasticity or hypotonia due to imbalance in muscle tone, posture disorders, uncontrolled movements and coordination disorders. Motor disorders are often accompanied by sensory, perceptual, cognitive, communication and behavioral problems, epilepsy and secondary musculoskeletal problems.

The European Cerebral Palsy Monitoring Group has divided SP into 3 classes: spastic, dyskinetic and ataxic types. The spastic type is divided into 2 types: unilateral spastic type SP, where one half of the body is affected, and bilateral spastic type SP, where both halves of the body are affected. Individuals with unilateral SP have low muscle tone, and increased muscle tone and increased reflexes are seen in the later stages. Due to antagonist muscle weakness, there is inability to perform quality lower extremity movements and maintain balance.

In the rehabilitation of individuals with CP, many treatment concepts with high evidence levels are used, such as action observation therapy, bimanual intensive training, treadmill training with partial body weight, hippotherapy, and target-oriented training, which are frequently studied in the literature. Constraint induced movement therapy is also one of the treatment methods that has been frequently used in recent years and has been proven to have positive effects in children with CP. Constraint induced movement therapy (CIMT) is a translational motor rehabilitation technique following CNS injury. The original concept involved restricting the unaffected extremity and forcing the affected extremity. Subsequent studies in humans included voluntary collective tasks or shaping practices with the affected extremity. As a result, CIMT has been reported to be effective in improving real-world arm use, motor function, and kinematic outcomes by causing changes in brain functions and structures. However, many changes have been made to the original protocol of CIMT over the years, including but not limited to the length of time for task practice, restriction, and the use of a transfer package.

CIMT has a very strong evidence base with studies. CIMT for the lower extremity is an intensive intervention method that has recently been reported with good results, based on a modification of the original CIMT for the upper extremity. The applicability of the protocol for the upper extremity may be due to the unilateral nature of the use of these extremities in most of our daily living activities. This may seem difficult for the lower extremities because humans are bipedal and this requires them to use both extremities simultaneously in daily living activities, especially walking. However, the positive results in the recovery of upper extremity motor function following CIMT and its contribution to improving the neurophysiological functions of the brain have convinced the neuroscience community to consider translating the technique to the lower extremities. CIMT also increases the expression of Growth-Associated Protein 43 (GAP 43) and the number of ΔFosB-positive cells, some of the biomarkers that play important roles in neural cell proliferation and neural and synaptic plasticity. Similarly, lower extremity movement is critical to brain health because decreased mobility results in decreased neural stem cell proliferation and altered cell turnover. Consequently, a lower extremity CIMT protocol is designed to include an intensive practice protocol with the predominantly affected extremity, shaping activities, transfer wrapping, and encouragement of increased use of the affected extremity. So far, there are several studies investigating the effects of lower extremity CIMT on walking parameters, balance, and motor function using different study designs, such as case reports, experimental studies, quasi-experimental studies, and randomized controlled trials. These studies reported that lower extremity CIMT improved walking speed, step length, motor function, functional mobility, balance, and kinematic outcomes.

Lower extremity constraint induced movement therapy has been applied to individuals with multiple sclerosis, stroke, subacute and chronic hemiparesis in recent years and positive results have been reported. However, there is no study in the literature regarding the application of this treatment method to the pediatric population. In order to address this gap in the literature, we planned to conduct this study to examine the possible effects of lower extremity constraint induced movement therapy on lower extremity functions, balance and gait parameters in individuals with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Cerebral Palsy by a Child Neurologist.
* Having been classified as Unilateral Cerebral Palsy according to SCPE.
* Being between the ages of 5-15,
* Being at levels I-II according to the Gross Motor Function Classification System
* Being at levels I-II according to the Communication Function Classification System
* Being able to stand up from sitting independently, even with the help of the upper extremity
* Being able to walk at least 10 m with or without an assistive device

Exclusion Criteria:

* Children who have had lower extremity orthopedic surgery within the last six months
* Children who have had lower extremity Botox injections within the last six months
* Those with rigid contractures involving lower extremity joints,
* Children with levels III-IV according to the Communication Functions Classification System
* Families and children who do not accept full participation in treatment

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Surface EMG | 6 weeks
  Electromyography is a method used to record and analyze myoelectric signals; it provides information about the transfer of the signals to the neuromuscular junction, the electrical activation of muscle cells in the motor unit, muscular contraction and relaxation strategies and activation time. sEMG measurements made on the individual's skin using superficial electrodes are frequently preferred for research purposes because they are non-invasive and painless. In sEMG application, electrodes are usually placed in the center of the muscle body for large superficial muscles and on the target muscle for small muscles. The maximal voluntary isometric contraction (MVIC) value of the muscles will be calculated and recorded with electromyographic evaluation in the individuals participating in the study. The results of the pre-evaluation and post-evaluation will be compared. The muscle groups to be evaluated within the scope of our study are M. Rectus Femoris and M. Gastrocnemius.

SECONDARY OUTCOMES:
Modified Tardieu Scale | 6 weeks
  It is a scale that evaluates the velocity-dependent part of spasticity recommended for use in the clinic. The resistance given to passive joint movement is evaluated between 0 and 5. The muscle reaction value (X) and muscle reaction angle (Y) are scored by measuring two different reaction angles at three different speeds.
  Muscle reaction values (X):
  (0) No resistance to passive movement
  1. There is slight resistance to passive movement but no "catch" sensation
  2. There is a "catch" sensation at a certain point
  3. Clonus lasting less than 10 seconds at a certain angle
  4. Clonus lasting more than 10 seconds at a certain angle
  5. The joint cannot be moved. Muscle Reaction Angle (Y) It will be measured according to the position where the muscle is minimally stretched. There are three different speeds (V1, V2, V3) and two different angular values (R1, R2).
  Scoring Criteria V1: as slow as possible V2: the speed of the extremities falling against gravity V3: as fast as possible
Gross Motor Function Measure (GMFM-88 Dimensions D and E) | 6 weeks
  GMFM is a standardized, valid and reliable scale that aims to determine capacity and change. It consists of five subsections: supine, prone and turning (A), sitting (B), crawling and kneeling (C), standing (D), walking, running and jumping (E). There are a total of 88 items in the subsections of GMFM. It is checked how much of each subsection the child has completed. Scoring is done according to a four-stage likert scale between 0-3. While the total score can be calculated, it is also possible to calculate each section on its own. Each section is converted into a percentage score within itself. Within the scope of our study, the evaluation will be made with the D and E sub-dimensions of GMFM-88 and percentage scores ranging from 0 to 100 will be calculated.
Selective Control Assessment of the Lower Extremity- SCALE | 6 weeks
  Normal selective voluntary motor control is the controlled performance of an isolated extremity movement without the occurrence of unwanted movements such as mirror-like movements and without the use of flexor and extensor patterns. The "Selective Control Assessment of the Lower Extremity- SCALE" test developed by Fowler et al. (21) in 2009 also evaluates the selectivity and quality of voluntary motor control of five regions (hip, knee, ankle, subtalar joint and toes) in the lower extremity. It has special definitions for each joint. According to the test scoring, the selectivity of the movement was defined as; 0=no movement
  1. voluntary movement can be initiated but cannot be performed in a fully controlled, selective and high-quality manner
  2. voluntary movement can be performed in a controlled, selective and high-quality manner.
  The highest SCALE score for each extremity is 10, and the total lower extremity selective motor control score is 20 points.
Observational Gait Analysis-OGS | 6 weeks
  It is an observational scale that rates the condition of the joints in the lower extremities according to the phases of walking. It was first used in the clinic by Koman et al. as the "Physician Rating Scale". OGS is an observational walking assessment that evaluates walking only in the sagittal plane. OGS, developed by Wren et al., evaluates the walking pattern with the items; knee position in the middle of the stance phase, first foot contact, foot contact in the middle of the stance phase, time of heel lift, rear foot in the middle of the stance phase, support area, use of assistive devices in walking. It measures from both the sagittal and frontal planes. The highest score for each extremity is 22. A high score indicates advanced walking skills. In this study, children will walk on a 6meter-long surface without devices, support or without support. Children of families who accept video recording will be videotaped during walking and the videos will be watched and OGS will be scored
Gross Motor Function Classification System | 6 weeks
  The gross motor function classification system (GMFCS), developed by Palisano et al. for children with cerebral palsy, is based on child-initiated movements, with emphasis on sitting, moving, and mobility. It consists of five levels.
  The general headings for each level are as follows.
  Level 1: Walks without restrictions. Level 2: Walks with restrictions. Level 3: Walks using hand-held mobility devices. Level 4: Self-mobility is limited. May use powered mobility. Level 5: Transported in a hand-propelled wheelchair.
Timed Up and Go Test | 6 weeks
  The Timed Up and Go Test is frequently used to assess functional mobility in adults. Williams et al. adapted the test for use in children, demonstrated the validity and reliability of the TUG in their study on healthy and disabled children, and reported that the TUG is a tool that can be used in children with special development and can measure changes in functional mobility over time. In a standard timed up and go test, the individual stands up from a chair, stands, walks 3 meters, and returns to the same chair, and the time between the command to stand and the individual sitting back in the chair is calculated.
Pediatric Balance Scale | 6 weeks
  It was developed by Franjoine et al. by modifying the adult "Berg Balance Scale". PBS has been shown to be valid and reliable in school-age children. It is a comprehensive and effective scale that evaluates balance in the following three dimensions: static balance, forward balance and functional movement transitions. The scale consists of 14 items including sitting balance, standing balance, sitting to standing/standing to sitting, transfers, taking steps, reaching forward with arm extended, reaching the ground, turning and placing foot on stool. Each item is rated from 0 to 4. 0 indicates inability to follow the instructions, while 4 indicates the ability to follow them without any difficulty. The lowest score that can be obtained from the scale is 0 and the highest score is 56, and as the score increases, it indicates advanced balance skills.
Gillette functional gait assessment questionnaire | 6 weeks
  The Gillette Functional Gait Assessment Questionnaire is a walking scale applied to families by asking questions, and is a questionnaire that evaluates the walking ability of neurologically affected children who can and cannot walk, in public and outside the community, on a scale of 0-10. 0 indicates that the child cannot take a step and walk; 10 indicates that the child can walk and run on all surfaces without assistance and can go up and down stairs. In this study, the Gillette functional gait assessment questionnaire will be administered to families of children with CP via face-to-face interviews.
Weight Transfer Test | 6 weeks
  Weight transfer to the affected and unaffected lower extremities of children with unilateral CP is planned to be done with two scales of the same brand. The measurement will be made while the children stand with their feet shoulder-width apart, each foot on a different scale. The amount of weight transferred to their healthy and affected lower extremities will be written in kilograms (kg), and the difference between the weight transfer of both lower extremities will be recorded in kg.
Pediatric Evaluation of Disability Inventory (PEDI) | 6 weeks
  It is a comprehensive clinical assessment tool that evaluates children's functional abilities and performance by asking the family. PEDI consists of three main sections under the subheadings of functional skills, caregiver assistance, and modifications. Each of these sections evaluates the areas of self-care, mobility, and social function. The functional skills section consists of 197 items and directly measures the child's functional abilities. In this section, the Self-Care subsection consists of 73 items, the Mobility subsection consists of 59 items, and the Social Functions subsection consists of 65 items. The child is given a score of 0; cannot do the items in this section and 1; can do them. At the end of each subsection, the scores of that section are added up and the Functional Skills Total Score is obtained by adding the scores of the subsections. The lowest score is 0 and the highest score is 197. As the score increases, the level of independence increases.
Goal Attaintment Scale (GAS) | 6 weeks
  It is widely used to evaluate the effects of individualized, targeted physiotherapy and rehabilitation programs for children with CP. In order to measure the effect of the treatment, child-specific goals are determined together with the family, child and specialists. Goals are graded on five levels between -2 and 2. Goals should be specific, measurable, achievable, resource-sensitive and timely (SMART).
  A value of "-2" indicates a value well below the desired goal, "-1" indicates a value below the desired goal, "0" indicates the desired goal, "1" indicates a success value above the desired goal, "2" indicates a success value well above the desired goal. It has a special calculation. For each target; the weighted score (Wi) is calculated according to the importance (i) and difficulty (d) scores (Wi=i X d).
Impact on Family Scale (IPFAM) | 6 weeks
  IPFAM was developed by Stein and Reissman in 1980 to measure the level of impact on families of children with chronic, systemic, or progressive diseases. IPFAM questions the family's financial support, the disruption caused by the condition in social relationships, coping power, general impact, and total impact levels. It was translated into Turkish by Bek et al. It was planned that the mothers or fathers of the children to be evaluated within the scope of our study would fill out this scale. The person who fills out the scale will be the person who is more involved in the child's care among the parents.
Communication Function Classification System (CFCS) | 6 weeks
  The Communication Function Classification System classifies the communication skills of children with CP at the level of activity and participation. It was developed as an analogue of the GMFCS and Manual Ability Classification System (MACS). The GMFCS used in classifying CP in the literature has also been found to be related to other classification systems such as MACS.
  Level 1: Effective giver and receiver with familiar and unfamiliar partners. The person can independently switch between giver and receiver roles with most people in most settings.
  Level 2: Effective but slow-paced giver and receiver with familiar and/or unfamiliar partners.
  Level 3: Effective giver and receiver with familiar partners. Level 4: Incompatible giver and/or receiver with familiar partners. The person's giver and receiver roles do not change continuously.
  Level 5: Rarely effective giver and receiver even with familiar partners. The person is a limited giver and receiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University Faculty of Health Sciences, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No